CLINICAL TRIAL: NCT07370298
Title: Developing and Testing a Digital Health Tool for INterseCtional Stigma Assessment and Reduction at Multiple Levels and mUltiple DimEnsions (INCLUDE) to Improve HIV Care in ART Centers in Nepal
Acronym: INCLUDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Possible (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institutes of Health (NIH) (NIH); National Center for AIDS and STD Control, Government of Nepal (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCLUDEPossible; 1R01TW012682 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV Care Loss to Followup; HIV Antiretroviral Therapy (ART) Adherence; HIV Stigma; Mental Health Conditions; Stigma; Intersectional Stigma; Gender Minority Individuals; Ethnic Minorities
Keywords: Stigma; Intersectional Stigma; HIV; HIV Care; Mental health conditions; Sexual and gender minorities; Ethnic minorities; digital health intervention
MeSH Terms: conditions — Social Stigma; Coitus

STUDY DESIGN:
Intervention Model Description: This study is a 9-month single-arm acceptability and feasibility pilot trial to test INCLUDE in diverse ART centers to prepare for a future cluster-randomized trial. We will conduct this study in four ART centers. The staff at these ART centers will be trained on the INCLUDE digital health tool and then incorporate it for the 9-month trial period into the ART center's daily operations. We will recruit 40 PLWHs, 10 from each ART center, who will use the tool as part of their care at the participating ART center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INCLUDE (Experimental): INterseCtional stigma assessment and reduction at multiple Levels and mUltiple DimEnsions (INCLUDE) is a new digital health tool with three components that can address the challenges in assessing, prioritizing, and addressing intersectional stigma in ART centers. The components include: 1) an assessment strategy that can be used during a clinic visit to collect both quantitative (i.e., ratings) and qualitative data (i.e., free text of client's perspectives) on intersectional stigma reported by people living with HIV (PLWH); 2) a dashboard that incorporates this stigma assessment data alongside routine clinical data (i.e., existing registry of clients in the ART center) so that ART centers can directly link stigma with care engagement, and also identify relevant stigma-reduction activities; and 3) a repository of evidence-based, culturally appropriate activities that can reduce stigma at the intrapersonal-, interpersonal-, and clinic-levels.
  Interventions: Behavioral: INCLUDE

INTERVENTIONS:
Behavioral: INCLUDE — INterseCtional stigma assessment and reduction at multiple Levels and mUltiple DimEnsions (INCLUDE) is a new digital health tool with three components that can address the challenges in assessing, prioritizing, and addressing intersectional stigma in ART centers. The components include: 1) an assessment strategy that can be used during a clinic visit to collect both quantitative (i.e., ratings) and qualitative data (i.e., free text of client's perspectives) on intersectional stigma reported by people living with HIV (PLWH); 2) a dashboard that incorporates this stigma assessment data alongside routine clinical data (i.e., existing registry of clients in the ART center) so that ART centers can directly link stigma with care engagement, and also identify relevant stigma-reduction activities; and 3) a repository of evidence-based, culturally appropriate activities that can reduce stigma at the intrapersonal-, interpersonal-, and clinic-levels.

SUMMARY:
People living with HIV (PLWH) have poor clinical outcomes when they are excluded from care due to intersectional stigma related to HIV, mental health (MH), and other dimensions. Recent studies and reviews have highlighted three major challenges in identifying and addressing intersectional stigma: a lack of stigma assessment strategies that are multi-dimensional and can be incorporated into routine clinical care, a lack of tailored stigma-reduction activities, and a lack of implementation of multi-level interventions. These gaps make it difficult to recognize and address intersectional stigma, leading to poor HIV care outcomes globally.

Digital health tools, co-designed with PLWH and healthcare workers (HCWs), have the potential to assist ART centers in addressing these challenges. Guided by the principles of human-centered design, our team has developed a digital tool with three components that can address the challenges in assessing, prioritizing, and addressing intersectional stigma in ART centers. The components include: 1) a dynamic assessment strategy that can be used during a clinic visit to collect both quantitative (i.e., ratings) and qualitative data (i.e., free text of client's perspectives) on stigma reported by PLWH; 2) a dashboard that incorporates this stigma assessment data alongside routine clinical data (i.e., existing registry of clients in the ART center) so that ART centers can directly link stigma with care engagement, and also identify relevant stigma-reduction activities; and 3) a repository of evidence-based, culturally appropriate activities that can reduce stigma at the intrapersonal-, interpersonal-, and clinic-levels.

The three components of the digital intervention are theoretically grounded and are based on prior studies and consultations with local partners. The study aims to assess the acceptability and feasibility of INCLUDE among clients, HCWs, and ART center leads in four ART centers. For this aim, we will conduct a pilot trial at four ART centers to assess the acceptability and feasibility of INCLUDE. If successful, this study will provide an intervention that can be incorporated into routine clinical practice to systematically identify and address intersectional stigma to improve HIV care, and can be tested in a cluster randomized trial with ART centers in Nepal and other regions that face similar challenges.

DETAILED DESCRIPTION:
Intersectional stigma is a pervasive barrier to care that disproportionately affects people living with HIV (PLWH) and leads to poor clinical outcomes. While the understanding of intersectional stigma is still evolving, it is based on intersectionality, a long-standing understanding that oppressive forces intersect to create and maintain inequity. A major challenge in achieving the 2025 UNAIDS 95-95-95 goals is the persistent intersectional stigma faced by PLWH who are marginalized and minoritized because of mental health (MH) problems, sexual and gender minority (SGM) status, race, and/or other dimensions. The relationship between these dimensions, intersectional stigma, and health outcomes is complex. Globally, key populations, who often face intersectional stigma, are more likely to become infected with HIV and less likely to initiate ART and achieve viral suppression. A 2021 systematic review found the prevalence of MH problems among PLWH to be 28-62%. Marginalized populations, who often face minority stress, are even more likely to report MH problems, which are associated with further (layered or intersecting) stigma and poor health outcomes. Therefore, addressing intersectional stigma is crucial for improving HIV outcomes and quality of life for PLWH.

The Nepali government's 2023 HIV report estimated there are 30,000 PLWH, 93% of whom are aware of their status, and 77% of those who were tested had initiated ART. However, only 54% of PLWH receiving ART had achieved viral load (VL) suppression, and this rate was low before the COVID pandemic as well: 47% in 2018 and 45% in 2019. These data highlight the importance of increasing HIV care engagement in Nepal. Although there is a lack of studies directly assessing intersectional stigma in Nepal, there is a high prevalence of stigma in the relevant dimensions of HIV, MH, SGM, and Dalit minoritized caste in Nepal. In a nationally representative 2022 study (N=927), stigma was highlighted as an important driver of poor care engagement and quality of life among Nepali PLWH. Prevalence of stigma and discrimination was high among SGMs (22-30%), with 19% reporting that health care workers (HCWs) were the source. Among PLWH who had interrupted ART in the last 12 months, 49% reported stigma as the main reason (e.g., fear of others finding out and poor treatment from HCWs). We have described the role of SGM stigma in worsening HIV outcomes in Nepal. The pervasiveness of MH stigma is well-documented in Nepal, including by our team, showing that HCWs have virtually no formal MH training and are often dismissive of people with MH problems. The importance of MH is further elevated because of the high rates of MH problems among PLWH both globally and in Nepal. Furthermore, because only 10% of people with MH problems receive any treatment at all, this allows MH problems to persist. As such, consistent with the goals of this study, there is an urgent need to develop and test interventions that address stigma from HIV, MH, and other dimensions among PLWH in low- and middle-income countries (LMICs) such as Nepal to achieve the goals of improved HIV outcomes. As the field of intersectional stigma grows, there are three major challenges that we seek to address with our intervention. There are multiple challenges in assessing intersectional stigma. There may not be a standard approach to measure something as complex as intersectional stigma, and several recommendations have emerged. First, assessments need to be multidimensional by capturing dynamic contributions from HIV, MH, and other dimensions such as SGM status and/or race (in Nepal, caste). Second, both quantitative and qualitative methods are necessary to capture the complex experiences of PLWH while also tracking trends at a systems-level. Third, assessments should be used routinely within regular clinical practice, both for long-term sustainability and to address the lack of routine stigma data from clinical settings. While assessments need to be multi-level (intrapersonal, interpersonal, organizational, and higher levels), they must incorporate the experiences of PLWH. Finally, assessments should be actionable by directly leading to stigma reduction interventions, and they need to be feasible to use within regular clinical practice.

Many interventions have been developed to address stigma, but they often focus on specific conditions (e.g., positive contact with a person with MH problems) and/or at a certain driver (e.g., HCW training to improve comfort and competency in working with SGM), and work at a specific level (e.g., client-level intervention to facilitate access to peers). However, because multidimensional intersectional stigma is driven by multiple drivers working at multiple levels, a major challenge is that stigma-reduction interventions are rarely tailored and customized to the stigma drivers, dimensions, and levels that affect individual clients. As an example, from our consultations in Nepal, if a racially minoritized transgender PLWH is feeling guilty about her decision to take hormones because they are exacerbating her anxiety and she is worried about being stigmatized and stereotyped for not having her emotions under control, this experience may worsen her internalized intersectional stigma from HIV, minority stress, SGM status, and having MH problems. In such a situation, implementing a clinic-wide policy aimed at just one dimension (e.g., developing SGM-friendly registration forms) or HCW training targeting one driver (e.g., dismantling negative SGM stereotypes) is unlikely to increase her engagement in care because these activities, while potentially helpful, are not tailored to her experience. Stigma-reduction activities are often sporadic and are rarely directly linked to specific concerns and experiences of PLWH. As such, there is a large gap in developing and testing interventions that can directly link PLWH concerns with the appropriate stigma-reduction activities.

A 2018 review of stigma-reduction activities for HIV, MH problems, and physical disabilities found that 99% of interventions were at intrapersonal or interpersonal levels rather than at organizational/structural levels. This is consistent with other reviews and recent calls for multi-level interventions. Because oppressive structural forces sustain intersectional stigma, interventions need to be multi-level and expand beyond the intrapersonal or interpersonal levels.

Digital health can facilitate novel approaches to address the aforementioned three challenges in assessing and addressing intersectional stigma using evidence-based, multi-level activities that are tailored to the dimensions and drivers that are most relevant to PLWH. We have developed a digital health tool INterseCtional stigma assessment and reduction at multiple Levels and mUltiple DimEnsions (INCLUDE) to improve HIV care in ART centers in Nepal. This tool was developed using a human-centered five-step design thinking approach, which is based on the principles of participatory co-design and can incorporate the perspectives of the end users and beneficiaries to develop tools that can help address the problems they face. This tool is designed to address the modifiable drivers of stigma and discrimination at multiple levels. At the organization-level, INCLUDE will routinely link stigma with poor HIV outcomes, enhancing its salience and importance. INCLUDE will provide ART centers with easily accessible stigma-reduction resources and strategies. At the HCW-level, it will facilitate positive contact with stigmatized individuals and deliver training targeting misconceptions and negative stereotypes. At the client level, INCLUDE will facilitate the identification of client-specific stigma drivers and provide a connection with peers who can provide support and acceptance. INCLUDE will provide access to evidence-based stress reduction strategies and referrals to providers who have been identified by local activists as being supportive and accepting of stigmatized individuals. By interrupting the pathways via which intersectional stigma reduces care engagement, we theorize that our multi-level intervention will improve HIV outcomes.

The overall goal of this study is to test a digital health tool INterseCtional stigma assessment and reduction at multiple Levels and mUltiple DimEnsions (INCLUDE) to improve HIV care in ART centers in Nepal. The specific objective of this study is to assess the acceptability and feasibility of INCLUDE among clients, HCWs, and ART center leads in four ART centers.

This pilot trial will use a single-arm design and will collect both quantitative and qualitative data to evaluate the tool's performance in real-world settings. Participants, including PLWH and HCWs, will be recruited from diverse ART centers, with a particular focus on ensuring representation from marginalized groups, such as Dalits and sexual and gender minorities (SGMs). The study will gather data through surveys, app usage analytics (paradata), in-depth interviews, and focus group discussions. This combination of data collection methods will provide a comprehensive understanding of how the tool is used and perceived, allowing for further refinement and potential scaling of INCLUDE.

ELIGIBILITY:
There are two groups of study participants: people living with HIV (PLWH) and healthcare workers (HCWs) in ART centers (clinics for HIV treatment) in Nepal.

1. Inclusion Criteria for PLWH:

   * PLWH with poor HIV outcomes (a. been in care for more than 6 months but with detectable VL; b. missed clinic visit by more than a month; and/or c. did not pick up medications for more than 2 weeks from the expected refill date);
   * age ≥18;
   * screening positive for having mental health conditions (with the Generalized Anxiety-7 and Patient Health Questionnaire-9 screening tools); and
   * living in the ART (Anti-Retroviral Therapy) center's catchment area with no plans to leave during the study period.
   * Sexual and Gender Minorities and/or Ethnic Minorities. Participants will be drawn randomly from this list, stratified by having additional stigma dimension(s) vs. not.
2. Exclusion Criteria for PLWH:

   * presence of significant cognitive problems/disability precluding participation
3. Inclusion Criteria for HCWs:

   * All HCWs of ART centers: HIV counselors, ART center leads, and other HCWs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability ratings | 9 months
  Acceptability of the INCLUDE tool among healthcare workers will be assessed via a quarterly survey. Ratings will be provided on a 5-point Likert scale ranging from 1 to 5, where higher scores indicate greater acceptability. The outcome will be reported as the proportion of healthcare workers with specific rating categories.
Acceptability of the INCLUDE tool | 4 and 9 months from baseline
  Acceptability among PLWHs will be measured by serial in-depth interviews (IDIs) to understand their perspectives and overall experience with the INCLUDE tool.
Rate of assessment app launch | 9 months
  We will use paradata collected passively from the INCLUDE tool to measure the rate of assessment app launch per client per quarter.
Assessment Duration | 9 months
  The mean duration, in minutes, required for clients to complete the INCLUDE assessment form. Duration is calculated using passively collected system paradata, tracking the time from assessment initiation to submission.
Frequency of assessment completion | 9 months
  The number of completed assessment forms submitted by clients in the INCLUDE tool.
Frequency of user-led early termination/non-completion | 9 months
  The number of times the platform launch was terminated early or not completed by users.
Frequency of application errors/crashes | 9 months
  Frequency of the INCLUDE tool displaying error messages or crashing while in use (proportion of all user encounters where an error message/application crash occurs)
Rate of client data completion in the INCLUDE tool's dashboard | 9 months
  The completion rate of client data in the INCLUDE tool's dashboard relative to the total number of clients registered.
Feasibility of the INCLUDE intervention | 4 and 9 months from baseline
  We will conduct serial in-depth interviews (IDIs) with people living with HIV to ask about them about the feasibility of using the INCLUDE tool.
Rate of INCLUDE conference meetings | 9 months
  The rate of INCLUDE conference meetings will be defined as the percentage of scheduled monthly conference meetings conducted. This data will be derived from the research staff logs.
Conference meeting time | 9 months
  We will measure the average length of time spent in each conference meeting from research staff logs.
Rate of stigma-reduction activity being recommended | 9 months
  We will measure the rate of at least one stigma-reduction activity being recommended in response to assessment data from each client, as recorded in the counselor form of the INCLUDE tool.
Implementation rate of recommended activities | 9 months
  We will track the implementation rate of recommended stigma reduction activities from past conference meetings.

CONTACTS AND LOCATIONS:
Overall Officials: Bibhav Acharya, MD, Principal Investigator — University of California, San Francisco; Sabitri Sapkota, PhD, Principal Investigator — Possible
Locations (1):
- Possible, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
We will publicly share the de-identified quantitative data by uploading in the National Institute of Mental Health (NIMH) Data Archive (NDA). For qualitative data, the documentation will include the structured notes.
Supporting Information: SAP, Analytic Code
Time Frame: IPD and supporting information will be available approximately 12 months following the end of the trial. IPD will be available to the research community in perpetuity.
Access Criteria: All shared data will be publicly accessible in the National Institute of Mental Health (NIMH) Data Archive (NDA).
URL: https://nda.nih.gov